CLINICAL TRIAL: NCT02705027
Title: Randomized, Controlled Comparison of Two Endoscopically Placed Nasojejunal Probes in Critically Ill Patients in Terms of Application Time and Technical Success
Brief Title: Comparison of Two Endoscopically Placed Nasojejunal Probes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Andrea Riphaus, PD Dr., Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 3967-11
Record Dates: First submitted 2016-02-18; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Investigation Time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Active Comparator): After randomization one half of the patients receive a Freka®-Trilumina probe, which is inserted in nasogastric route an then "pushed " using a small forceps which is inserted through the endoscope into the small intestine.
  Interventions: Device: Freka®-Trilumina versus Freka®-EasyIn
- Freka®-EasyIn (Experimental): The other half of the patients will receive a Freka®-EasyIn probe which is directly placed in the small intestine inserted over the endoscope, after endoscopy was initially pushed - as far as possible - into the small intestine.
  Interventions: Device: Freka®-Trilumina versus Freka®-EasyIn

INTERVENTIONS:
Device: Freka®-Trilumina versus Freka®-EasyIn — Direct placement of probe via endoscope

SUMMARY:
A direct application of jejunal tube feeding is necessary especially in patients with gastroparesis due of existing diabetes mellitus, postoperative or severe underlying disease. Since the jejunal tube feedings, the secretion of gastric juice can be increased, the use of probes that allow both: jejunal nutrition, as well as a gastric outflow of secretions are beneficial.

While in a randomized trial of Schwab et al. it could be shown that the use of Freka-Trilumina® compared to Dobbhoff probe by so-called drag technique is significantly faster there are currently no comparative data to use the Easy-In® probe subsequently developed , which is directly introduced through the working channel of the endoscope, and thus shortening the procedure time.

DETAILED DESCRIPTION:
The use of probes nasojejunal has increasingly become important especially in critically ill patients because of the beneficial effect in patients e.g. with necrotizing pancreatitis, according trauma or major surgical procedures.

A direct application of jejunal tube feeding is necessary especially in patients with gastroparesis due of existing diabetes mellitus, postoperative or severe underlying disease. Since the jejunal tube feedings, the secretion of gastric juice can be increased, the use of probes that allow both: jejunal nutrition, as well as a gastric outflow of secretions are beneficial.

While in a randomized trial of Schwab et al. it could be shown that the use of Freka-Trilumina® compared to Dobbhoff probe by so-called drag technique is significantly faster there are currently no comparative data to use the Easy-In® probe subsequently developed , which is directly introduced through the working channel of the endoscope, and thus shortening the procedure time.

In the presented study should be investigated to what extent the use of imported directly via the working channel Easy-Inn® probe, application time and thus the investigation period may be shortened compared to the usual nasojenunal probes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical indication for enteral feeding via naso-jejunal probe

Exclusion Criteria:

* Lack of consent of the patient or their relatives (in intubated and mechanically ventilated patients in intensive care)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Examination time for the probe system | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - PD Dr. Andrea Riphaus, Hanover
  - Klinikum Agness Karll Laatzen, Laatzen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwab D, Muhldorfer S, Nusko G, Radespiel-Troger M, Hahn EG, Strauss R. Endoscopic placement of nasojejunal tubes: a randomized, controlled, prospective trial comparing suitability and technical success for two different tubes. Gastrointest Endosc. 2002 Dec;56(6):858-63. doi: 10.1067/mge.2002.129870. PMID 12447298